CLINICAL TRIAL: NCT03144206
Title: Randomized Pilot Study Evaluating Hyperbaric Oxygen Therapy Following Management of Soft Tissue Sarcoma With Neo-adjuvant Radiation and Surgical Resection
Brief Title: Hyperbaric Oxygen Therapy for Soft Tissue Sarcoma Pilot Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00065596
Record Dates: First submitted 2017-05-03; First posted 2017-05-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Sarcoma; Hyperbaric Oxygen Therapy
MeSH Terms: conditions — Sarcoma | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric Oxygen Group (Experimental): Patients will receive Hyperbaric Oxygen treatments in the immediate postoperative period
  Interventions: Drug: Hyperbaric oxygen
- Standard of Care Group (No Intervention): Patients will not receive Hyperbaric Oxygen treatments in the immediate postoperative period

INTERVENTIONS:
Drug: Hyperbaric oxygen — Patients with soft tissue sarcomas will receive HBOT treatment in the immediate postoperative period
  Arms: Hyperbaric Oxygen Group

SUMMARY:
A parallel-group randomized pilot trial at a single institution (Duke University) on the effect of postoperative hyperbaric oxygen therapy on wound healing in patients with soft tissue sarcoma undergoing surgical resection with neo-adjuvant radiation therapy.. Participants will be allocated to either the treatment group (HBOT) or control (standard of care) by computer-generated randomization, stratified by tumor size (≤10cm and >10cm). An unequal randomization of 2:1 will be utilized to provide experience prescribing HBOT to more patients.

DETAILED DESCRIPTION:
Patients with a primary diagnosis of soft tissue sarcoma of the lower extremities undergoing treatment with neo-adjuvant radiation therapy and surgical resection will be screened for eligibility. All participants will receive pre-operative radiation treatment per standard of care and will undergo surgical excision as planned and performed by one of the surgical oncologists at our center. Participants randomized to the treatment group will be scheduled for 7-10 HBO treatments within 7-10 days of surgery. All participants will be scheduled for follow-up visits with their surgical oncologist at the following post-operative time points: 3, 6, 12, and 24-weeks (+/- 14 days). Follow up for the purposes of this study will continue up to 6 months from the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females within the ages of 18-85
2. Diagnosis of soft tissue sarcoma that has been histologically confirmed by an approved reference pathologist
3. Sarcoma of lower extremity location
4. Treatment plan that includes neo-adjuvant radiation therapy followed by surgical resection
5. Expected primary wound closure performed at the time at surgery
6. Any disease stage
7. Any tumor grade
8. Any histologic subtype
9. First or recurrent presentations
10. No vascular invasion or resection/repair/reconstruction that results in decreased perfusion of the extremity
11. No history of radiation therapy to the tumor and/or surgical area prior to the current treatment being studied
12. Must be able to comply with follow up visits
13. Must be able to provide own consent

Exclusion Criteria:

1. Patients under the age of 18, or over the age of 85.
2. Treatment plan that doesn't include neo-adjuvant radiation and surgical excision
3. Sarcoma location other than lower extremity
4. History of radiation therapy to the tumor and/or surgical area prior to the current treatment being studied
5. High dose steroid therapy (defined as >5mg prednisone, or equivalent, daily)
6. Active treatment with chemotherapy
7. Inability of the patient to provide informed consent (i.e. dementia, cognitive impairment, non-English speakers)
8. Plan for post operative radiation therapy
9. Vascular invasion or resection/repair/reconstruction that results in decreased perfusion of the extremity
10. Vascular disease resulting in clinically apparent compromise in blood flow to the treatment extremity (i.e. peripheral vascular disease with diminished pulses, venous insufficiency with clinical evidence of vascular congestion)
11. Actively uncontrolled diabetes mellitus (documentation of history of diabetes mellitus with A1c>8)
12. Active deep vein thrombosis in the treatment extremity
13. Inability to comply with follow up visits
14. Pregnant females (women of childbearing potential must have a negative serum pregnancy test prior to enrollment)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Screening
  The proportion of eligible patients who enroll in this study, as indicated by the screening log.
Hyperbaric Treatment Completion Rate | 24 weeks postoperatively
  The proportion of prescribed hyperbaric oxygen treatments that are completed, which will be recorded in the appointment log.
Wound Assessment Form Completion Rate | 24 weeks postoperatively
  The number of completed Wound Assessment Forms per participant divided by the total number of follow-up visits per participant.
Participant Assessment Form Completion Rate | 24 weeks postoperatively
  Number of completed Participant Assessment Forms per participant divided by the number of total follow-up visits per participant.
patient reported study strengths and weaknesses | 24 weeks postoperatively
  The Patient Feedback Survey will be given to all participants at their final study-related visit in order to collect qualitative and quantitative data on patient reported study strengths and weaknesses.
barriers to compliance with study procedures | 24 weeks postoperatively
  The Patient Feedback Survey will be given to all participants at their final study-related visit in order to collect qualitative and quantitative data on patient reported barriers to compliance with study procedures

SECONDARY OUTCOMES:
Frequency of surgical site infections or periprosthetic infections | 24 weeks postoperatively
  the number of participants with ≥ 1 completed Wound Assessment Form documenting infection or treatment for infection around the wound area at any follow-up visit.
frequency of wound complications that result in a secondary procedure | 24 weeks postoperatively
  the number of participants with ≥ 1 completed Wound Assessment Form that documents reoperation or any other invasive procedure after primary resection with any wound complication as the indication for the procedure.
Wound Severity | 24 weeks postoperatively
  Variability in clinical evaluations of wound severity will be determined by the Bates-Jensen Wound Assessment score recorded in the Wound Assessment Form.
Frequency of delayed wound healing | 24 weeks postoperatively
  The frequency of delayed wound healing will be determined by the number of participants with of ≥ 1 completed Wound Assessment Form documenting ≥ 1 clinical indication of a wound complication at any follow-up visit.
Variability in Patient Reported Quality of Life | 24 weeks postoperatively
  Variability in patient reported outcome data pertaining to quality of life will be determined by the ESAS-SM score alone at baseline and by the ESAS-SM and WOUND-Q: Life Impact scores recorded in the Participant Assessment Form at all follow-up visits.
Variability in Patient Reported Wound Assessments | 24 weeks postoperatively
  Variability in patient reported outcome data pertaining to wound assessments will be determined by the WOUND-Q: Wound Characterization score recorded in the Participant Assessment Form at all follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: William Eward, MD, DVM, Principal Investigator — Duke Health
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No